CLINICAL TRIAL: NCT00646763
Title: A Phase II Single Institution Randomized Study Comparing Cytokine Administration Sites for Mobilization of Peripheral Hematopoietic Progenitor Cells for Patients Undergoing Autologous Hematopoietic Progenitor Cell Transplant
Brief Title: A Randomized Study of the Site for Growth Factor Injection for Patients Undergoing Autologous Stem Cell Transplantation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Accrual goal met
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Edmund Waller, Principal Investigator, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00007445; 7445 (Other: Other)
Record Dates: First submitted 2008-03-25; First posted 2008-03-28 (Estimated); Results first posted 2012-05-11 (Estimated); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Cytokines
MeSH Terms: interventions — Granulocyte Colony-Stimulating Factor; Filgrastim; sargramostim; Intercellular Signaling Peptides and Proteins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Abdomen (Active Comparator): These subjects will have their cytokine injections administered only to their abdomen.
  Interventions: Drug: G-CSF and GMCSF administered at abdomen
- Extremities (Active Comparator): The extremity arm will have their injections administered to their upper and/or lower extremities.
  Interventions: Drug: G-CSF, GM-CSF administered at extremities

INTERVENTIONS:
Drug: G-CSF, GM-CSF administered at extremities — Injection site Extremities: G-CSF injections will commence on the day after completion of mobilization chemotherapy, at least 24 hours after completion of the last chemotherapy dose. On the seventh day of cytokine administration, GMCSF injections will be started, and patients will maintain a twice daily schedule of G-CSF/GM-CSF until stem cell collection is complete.
  Other Names: Neupogen, Leukine, growth factors
  Arms: Extremities
Drug: G-CSF and GMCSF administered at abdomen — Injection site Abdomen: G-CSF injections will commence on the day after completion of mobilization chemotherapy, at least 24 hours after completion of the last chemotherapy dose. On the seventh day of cytokine administration, GMCSF injections will be started, and patients will maintain a BID schedule of G-CSF/GM-CSF until stem cell collection is complete.
  Other Names: Neupogen, Leukine, growth factors
  Arms: Abdomen

SUMMARY:
The purpose of this study is to determine whether or not the injection site of cytokines, or growth factors, has an effect on peripheral blood stem cell collection.

DETAILED DESCRIPTION:
The purpose of this study is to determine the preferred injection site for G-CSF and GM-CSF, which are cytokines, or growth factors. The doctor may also choose to use these growth factors in combination with chemotherapy to increase the number of stem cells in the blood. Both options are established and are effective in increasing the number of stem cells in the blood.

Patients will receive one shot under the skin twice a day for approximately 12-15 days after receiving chemotherapy through the time your cells are being collected. Patients will be randomly assigned to receive growth factors administered either to their abdomen or to their extremities. Both shots will always be given either in the abdomen or in the extremities.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing autologous peripheral blood stem cell transplant (PBSC) for relapsed/refractory Hodgkin's disease, non-Hodgkin's lymphoma, or patients with myeloma. All patients must meet criteria for transplantation.

Exclusion Criteria:

* Patients with active, invasive/systemic fungal infection.
* Patients who are pregnant or lactating females.
* Patients with active CNS malignant disease or life expectancy limited by diseases other than the disease for which the patient is being transplanted.
* Also, patients cannot have known hypersensitivity to either G-CSF or GM-CSF.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2008-04; Primary Completion 2009-09 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edmund Waller, MD, Principal Investigator — Emory University Winship Cancer Institute
Locations (1):
- Emory University Winship Cancer Institute, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Abdomen | Extremities
Started | 18 | 17
Completed | 18 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Abdomen | Extremities | Total
Number analyzed (Participants) | 18 | 17 | 35
Age, Customized [Mean (Standard Deviation); unit: Mean] | 53 (13.76) | 52 (17.02) | 53 (15.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 7 | 17
  Male | 8 | 10 | 18
Region of Enrollment [Number; unit: participants]
  United States | 18 | 17 | 35
Disease type [Number; unit: participants]
  Lymphoma | 4 | 6 | 10
  Myeloma | 14 | 11 | 25

OUTCOME MEASURES:

1. Primary Outcome: The Total Number of CD34+ Cells Collected.
Time Frame: 4 days
Population: Patients at our institution between the ages of 18 and 70 years old with relapsed or refractory Hodgkin's disease, non-Hodgkin's lymphoma, or mutiple myelomawhowere scheduled for an autologous HSCTwere eligible to participate in the study.
Measure: Mean (Standard Deviation); unit: cells per Kg
Arm/Group | Abdomen | Extremities
Number analyzed (Participants) | 18 | 17
cells per Kg | 9,150,000 (4,700,000) | 9,850,000 (4,970,000)

2. Secondary Outcome: Total Number of Days of Apheresis
Description: the number of days of apheresis required to collect target numbers of CD34+ cells.
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Abdomen | Extremities
Number analyzed (Participants) | 18 | 17
days | 2.18 (1.01) | 2.00 (0.97)

3. Primary Outcome: Number of Participants for Whom Target Number of CD34+ Cells Were Collected.
Description: Target numbers of CD34+ cells for a single autologous transplant are typically at least 5.0 * 10^6 cells/kg, a cell dose that consistently results in rapid cell engraftment
Time Frame: 7 days
Measure: Number; unit: participants
Arm/Group | Abdomen | Extremities
Number analyzed (Participants) | 18 | 17
participants | 10 | 9

ADVERSE EVENTS:
Arm/Group | Abdomen | Extremities
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/17
Other Adverse Events (participants affected / at risk) | 18/18 | 17/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abdomen (N=18) | Extremities (N=17)
Bone Pain (Musculoskeletal and connective tissue disorders) | 18 | 17
Redness at the injection site (Skin and subcutaneous tissue disorders) | 18 | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No